CLINICAL TRIAL: NCT04902105
Title: A Phase 1, Open-Label, Fixed Sequence, Drug-Drug Interaction Study to Evaluate the Effect of Inhibition of Uridine 5'-Diphosphate-glucuronosyltransferases (UGTs) on the Pharmacokinetics of Ecopipam Tablets and Its Active Metabolite (EBS-101-40853) in Healthy Subjects
Brief Title: Drug-Drug Interaction Study to Evaluate the Effect of Inhibition of UGTs on the PK of Ecopipam and Its Active Metabolite
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Emalex Biosciences Inc. (Industry)
Collaborators: Syneos Health (Other); Nuventra, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: EBS-101-HV-102
Record Dates: First submitted 2021-05-20; First posted 2021-05-26 (Actual); Last update posted 2021-07-22 (Actual); Status verified 2021-07

CONDITIONS: Drug Interaction
MeSH Terms: interventions — Mefenamic Acid

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Cohort A (Other): Ecopipam HCL - 2 doses of 200mg
  Mefenamic acid 250mg Q6H for 7 days
  Interventions: Drug: ecopipam HCL; Drug: Mefenamic acid
- Cohort B (Other): Ecopipam HCL - 2 doses of 200mg
  Divalproex acid 1250mg QD for 10 days
  Interventions: Drug: ecopipam HCL; Drug: Divalproex Sodium ER

INTERVENTIONS:
Drug: ecopipam HCL — oral tablets
Drug: Mefenamic acid — oral capsules
  Arms: Cohort A
Drug: Divalproex Sodium ER — oral tablets
  Arms: Cohort B

SUMMARY:
This is a single center, open-label, fixed sequence, drug-drug interaction (DDI) study in healthy subjects.

DETAILED DESCRIPTION:
Following a 28-day Screening period, eligible subjects will enter the clinical research unit (CRU) and will be enrolled into either Cohort A or B. Subjects in both cohorts will receive a single dose of ecopipam on Day 1. On Day 7, subjects will begin taking a UGT inhibitor according to their assigned cohort. Subjects in Cohort A will receive mefenamic acid 250 mg every 6 hours for 7 days, while subjects in Cohort B will receive divalproex sodium ER 1250 mg once a day for 10 days. A single oral dose of ecopipam will also be administered to Cohort A on Day 7, 1 hour after the first dose of mefenamic acid, and to Cohort B on Day 10, 1 hour after administration of divalproex sodium ER. Subjects in Cohort A will continue taking mefenamic acid through the evening of Day 13 and will remain in the CRU until discharged on Day 14/ET. Subjects in Cohort B will continue taking divalproex sodium ER through Day 16 and will remain in the CRU until discharge on Day 17/ET.

ELIGIBILITY:
Inclusion Criteria:

* Male subjects or female subjects of non-childbearing potential
* ≥18 and ≤55 years of age at the time of consent
* BMI >18.5 and <30 kg/m2 and a weight of ≥50 kg
* Sexually active males must use a double barrier method of contraception during the study and for at least 90 days after the last dose of study drug
* Male subjects must be willing not to donate sperm until 90 days following the last study drug administration

Exclusion Criteria:

* Personal or family History of significant medical illness
* Clinically significant abnormalities on screening tests/exams
* History of or significant risk of committing suicide
* Donation of plasma within 7 days prior to dosing
* Donation or significant loss of blood within 30 days prior to the first dosing
* Major surgery within 3 months or minor surgery within 1 month prior to admission
* Use of prohibited prescription, over-the-counter medications or natural health products
* Alcohol-based products 24 hours prior to admission
* Female subjects who are currently pregnant or lactating
* Use of tobacco or nicotine products within 3 months prior to Screening
* Significant alcohol consumption
* History of drug abuse within the previous 2 years, or a positive drug screen
* History of allergy to study medications
* Not suitable for study in the opinion of the Principal Investigator

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2021-05-13 (Actual); Primary Completion 2021-07-06 (Actual); Study Completion 2021-07-06 (Actual)

PRIMARY OUTCOMES:
Cmax of ecopipam in the presence of mefenamic acid | Up to Day 16
  Up to 35 blood samples will be collected at the indicated time points for pharmacokinetic analysis
Cmax of ecopipam in the absence of mefenamic acid | Up to Day 16
  Up to 35 blood samples will be collected at the indicated time points for pharmacokinetic analysis
Cmax of ecopipam in the presence of divalproex sodium ER | Up to Day 16
  Up to 35 blood samples will be collected at the indicated time points for pharmacokinetic analysis
Cmax of ecopipam in the absence of divalproex sodium ER | Up to Day 16
  Up to 35 blood samples will be collected at the indicated time points for pharmacokinetic analysis
AUCinf of ecopipam in the presence of mefenamic acid | Up to Day 16
  Up to 35 blood samples will be collected at the indicated time points for pharmacokinetic analysis
AUCinf of ecopipam in the absence of mefenamic acid | Up to Day 16
  Up to 35 blood samples will be collected at the indicated time points for pharmacokinetic analysis
AUCinf of ecopipam in the presence of divalproex sodium ER | Up to Day 16
  Up to 35 blood samples will be collected at the indicated time points for pharmacokinetic analysis
AUCinf of ecopipam in the absence of divalproex sodium ER | Up to Day 16
  Up to 35 blood samples will be collected at the indicated time points for pharmacokinetic analysis
AUC0-143 of ecopipam in the presence of mefenamic acid | Up to Day 16
  Up to 35 blood samples will be collected at the indicated time points for pharmacokinetic analysis
AUC0-143 of ecopipam in the absence of mefenamic acid | Up to Day 16
  Up to 35 blood samples will be collected at the indicated time points for pharmacokinetic analysis
AUC0-143 of ecopipam in the presence of divalproex sodium ER | Up to Day 16
  Up to 35 blood samples will be collected at the indicated time points for pharmacokinetic analysis
AUC0-143 of ecopipam in the absence of divalproex sodium ER | Up to Day 16
  Up to 35 blood samples will be collected at the indicated time points for pharmacokinetic analysis

SECONDARY OUTCOMES:
Cmax of EBS-101-40853 | Up to Day 16
  Up to 35 blood samples will be collected at the indicated time points for pharmacokinetic analysis
AUCinf of EBS-101-40853 | Up to Day 16
  Up to 35 blood samples will be collected at the indicated time points for pharmacokinetic analysis
AUC0-143 of EBS-101-40853 | Up to Day 16
  Up to 35 blood samples will be collected at the indicated time points for pharmacokinetic analysis
Cmax of mefenamic acid | Up to Day 16
  Up to 15 blood samples will be collected at the indicated time points for pharmacokinetic analysis
Tmax of mefenamic acid | Up to Day 16
  Up to 15 blood samples will be collected at the indicated time points for pharmacokinetic analysis
AUCtau of mefenamic acid | Up to Day 16
  Up to 15 blood samples will be collected at the indicated time points for pharmacokinetic analysis
t½ of mefenamic acid | Up to Day 16
  Up to 15 blood samples will be collected at the indicated time points for pharmacokinetic analysis
Cmax of VPA | Up to Day 16
  Up to 19 blood samples will be collected at the indicated time points for pharmacokinetic analysis
Tmax of VPA | Up to Day 16
  Up to 19 blood samples will be collected at the indicated time points for pharmacokinetic analysis
AUCtau of VPA | Up to Day 16
  Up to 19 blood samples will be collected at the indicated time points for pharmacokinetic analysis
Safety and tolerability as demonstrated by MOAA/S | Up to Day 17
  Safety and tolerability measures will be recorded at the indicated timepoints.
Safety and tolerability as demonstrated by C-SSRS | Up to Day 17
  Safety and tolerability measures will be recorded at the indicated timepoints.
Safety and tolerability as demonstrated by concomitant medications | Up to Day 42
  Safety and tolerability measures will be recorded at the indicated timepoints.
AEs with relatedness associated with mefenamic acid | Up to Day 42
  Subjects will be continually monitored for adverse events
AEs with relatedness associated with divalproex sodium ER | Up to Day 42
  Subjects will be continually monitored for adverse events
AEs with relatedness associated with ecopipam | Up to Day 42
  Subjects will be continually monitored for adverse events
Absolute values of white blood cell (WBC) count (K/Ul) | Up to Day 17
  Blood samples will be collected for the assessment of hematology parameters.
Absolute values of neutrophils, lymphocytes, monocytes, eosinophils, and basophils (10E3/uL) | Up to Day 17
  Blood samples will be collected for the assessment of hematology parameters.
Absolute values of platelets (K/uL) | Up to Day 17
  Blood samples will be collected for the assessment of hematology parameters.
Absolute values of hematocrit (%) | Up to Day 17
  Blood samples will be collected for the assessment of hematology parameters.
Absolute values of hemoglobin (g/dL) | Up to Day 17
  Blood samples will be collected for the assessment of hematology parameters.
Absolute values of Red blood cell (RBC) count (M/uL) | Up to Day 17
  Blood samples will be collected for the assessment of hematology parameters.
Absolute values of blood sodium, magnesium, urea, phosphorus, potassium, and chloride (mg/dL) | Up to Day 17
  Blood samples will be collected for the assessment of clinical chemistry parameters.
Absolute values of creatinine, calcium, glucose, and direct and total bilirubin (mg/dL) | Up to Day 17
  Blood samples will be collected for the assessment of clinical chemistry parameters.
Absolute values of albumin and total protein (g/dL) | Up to Day 17
  Blood samples will be collected for the assessment of clinical chemistry parameters.
Absolute values of alanine aminotransferase (ALT), aspartate aminotransferase (AST), alkaline phosphatase (ALP), gamma glutamyl transferase (GGT), and creatinine phosphokinase (CPK) | Up to Day 17
  Blood samples will be collected for the assessment of clinical chemistry parameters.
Absolute values of urine specific gravity | Up to Day 17
  Urine samples will be collected for the assessment of urine parameters.
Absolute values of urine pH | Up to Day 17
  Urine samples will be collected for the assessment of urine parameters.
Absolute values of urine glucose | Up to Day 17
  Urine samples will be collected for the assessment of urine parameters.
Absolute values of urine protein | Up to Day 17
  Urine samples will be collected for the assessment of urine parameters.
Absolute values of urine blood | Up to Day 17
  Urine samples will be collected for the assessment of urine parameters.
Absolute values of urine ketones | Up to Day 17
  Urine samples will be collected for the assessment of urine parameters.
Absolute values of urine bilirubin, urobilinogen, and nitrite | Up to Day 17
  Urine samples will be collected for the assessment of urine parameters.
Absolute values of urine leukocytes by dipstick | Up to Day 17
  Urine samples will be collected for the assessment of urine parameters.
Change from Day -1 to Day of Discharge in white blood cell (WBC) count (K/Ul) | Up to Day 17
  Blood samples will be collected for the assessment of hematology parameters.
Change from Day -1 to Day of Discharge in neutrophils, lymphocytes, monocytes, eosinophils, and basophils (10E3/uL) | Up to Day 17
  Blood samples will be collected for the assessment of hematology parameters.
Change from Day -1 to Day of Discharge in platelets (K/uL) | Up to Day 17
  Blood samples will be collected for the assessment of hematology parameters.
Change from Day -1 to Day of Discharge in hematocrit (%) | Up to Day 17
  Blood samples will be collected for the assessment of hematology parameters.
Change from Day -1 to Day of Discharge in hemoglobin (g/dL) | Up to Day 17
  Blood samples will be collected for the assessment of hematology parameters.
Change from Day -1 to Day of Discharge in Red blood cell (RBC) count (M/uL) | Up to Day 17
  Blood samples will be collected for the assessment of hematology parameters.
Change from Day -1 to Day of Discharge in blood sodium, magnesium, urea, phosphorus, potassium, and chloride (mg/dL) | Up to Day 17
  Blood samples will be collected for the assessment of clinical chemistry parameters.
Change from Day -1 to Day of Discharge in creatinine, calcium, glucose, and direct and total bilirubin (mg/dL) | Up to Day 17
  Blood samples will be collected for the assessment of clinical chemistry parameters.
Change from Day -1 to Day of Discharge in albumin and total protein (g/dL) | Up to Day 17
  Blood samples will be collected for the assessment of clinical chemistry parameters.
Change from Day -1 to Day of Discharge in alanine aminotransferase (ALT), aspartate aminotransferase (AST), alkaline phosphatase (ALP), gamma glutamyl transferase (GGT), and creatinine phosphokinase (CPK) (U/L) | Up to Day 17
  Blood samples will be collected for the assessment of clinical chemistry parameters.
Change from Day -1 to Day of Discharge in urine specific gravity | Up to Day 17
  Urine samples will be collected for the assessment of urine parameters.
Change from Day -1 to Day of Discharge in urine pH | Up to Day 17
  Urine samples will be collected for the assessment of urine parameters.
Change from Day -1 to Day of Discharge in urine glucose | Up to Day 17
  Urine samples will be collected for the assessment of urine parameters.
Change from Day -1 to Day of Discharge in urine protein | Up to Day 17
  Urine samples will be collected for the assessment of urine parameters.
Change from Day -1 to Day of Discharge in urine blood | Up to Day 17
  Urine samples will be collected for the assessment of urine parameters.
Change from Day -1 to Day of Discharge in urine ketones | Up to Day 17
  Urine samples will be collected for the assessment of urine parameters.
Change from Day -1 to Day of Discharge in urine bilirubin, urobilinogen, and nitrite (Milligrams per deciliter) | Up to Day 17
  Urine samples will be collected for the assessment of urine parameters.
Change from Day -1 to Day of Discharge in urine leukocytes by dipstick | Up to Day 17
  Urine samples will be collected for the assessment of urine parameters.
Change from Day 6 to Day of Discharge in alanine aminotransferase (ALT) and aspartate aminotransferase (AST) (U/L) | Up to Day 17
  Blood samples will be collected for the assessment of clinical chemistry parameters.
Absolute values of electrocardiogram (ECG) parameters: PR, QRS, QT, and QT interval corrected for heart rate using Fridericia's formula (QTcF) (Milliseconds) | Up to Day 10
  Twelve-lead ECGs will be obtained with the participant in a supine position after a rest of at least 5 minutes using an automated ECG machine. PR, QRS, QT, and QTcF intervals will be measured.
Change from pre-dose for the respective day in ECG parameters: PR, QRS, QT, and QTcF (Milliseconds) | Up to Day 10
  Twelve-lead ECGs will be obtained with the participant in a supine position after a rest of at least 5 minutes using an automated ECG machine. PR, QRS, QT, and QTcF intervals will be measured.
Absolute values of oral temperature (degrees Celsius) | Up to Day 17
  Temperature will be assessed as part of vital signs.
Change from pre-dose for the respective day in oral temperature (degrees Celsius) | Up to Day 17
  Temperature will be assessed as part of vital signs.
Absolute values of heart rate (beats/minute) | Up to Day 17
  Heart rate will be assessed as part of vital signs.
Change from pre-dose for the respective day in heart rate (beats/minute) | Up to Day 17
  Heart rate will be assessed as part of vital signs.
Absolute values of respiratory rate (breaths/minute) | Up to Day 17
  Respiratory rate will be assessed as part of vital signs.
Change from pre-dose for the respective day in respiratory rate (breaths/minute) | Up to Day 17
  Respiratory rate will be assessed as part of vital signs.
Absolute values of systolic blood pressure (SBP) and diastolic blood pressure (DBP) (mmHG) | Up to Day 17
  Blood pressure will be assessed as part of vital signs.
Change from pre-dose for the respective day in SBP and DBP (mmHG) | Up to Day 17
  Blood pressure will be assessed as part of vital signs.

CONTACTS AND LOCATIONS:
Locations (1):
- Syneos Health Clinical Research Services, LLC., Miami, Florida, United States